CLINICAL TRIAL: NCT04515420
Title: The Influence of Noradrenaline Infusion on Coagulation and Fibrinolysis in Patients With Isolated Severe Brain Injury
Brief Title: The Influence of Noradrenaline on Coagulation and Fibrinolysis in Severe Isolated Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Adela Stecher, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: 123456
Record Dates: First submitted 2020-08-07; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Brain Injuries, Traumatic; Coagulopathy; Coagulation Defect; Acquired; Coagulation Defect; Bleeding; Fibrinolytic Hemorrhage, Acquired
Keywords: noradrenaline; thrombin generation; activation of coagulation; fibrinolysis; coagulation inhibition
MeSH Terms: conditions — Brain Injuries, Traumatic; Hemostatic Disorders; Hemorrhage | interventions — Norepinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Group A for patients that will need an infusion of NA solution to meet the desired CPP.
  Group A will be further divided into three sub-groups: A1 for patients that will receive NA in the dose of 0.06-0.12 μg/kg/min, A2 for patients that will receive a dose of 0.13-0.2 μg/kg/min, and A3 for patients that will receive a dose of NA > 0.2 μg/kg/min.
  Interventions: Drug: noradrenaline
- Group B: Group B for patients that will not receive NA infusion.

INTERVENTIONS:
Drug: noradrenaline — noradrenaline infusion
  Groups: Group A

SUMMARY:
Aim of the study

The investigators aim to establish:

* Whether noradrenaline (NA) infusion has a significant effect on coagulation and fibrinolysis in patients with severe traumatic brain injury (TBI).
* Whether disruption of haemostasis can be recorded with a computerized tomography (CT) scan.
* Whether there is a significant difference between the values of haemostasis parameters in the internal jugular vein and the radialis artery.

The hypotheses

1. In the early stage of treatment (1-3 hours), an increased formation of thrombin occurs in patients with severe isolated TBI that are treated with NA; consequently, platelet use increases in comparison with patients who don't need NA, as do coagulation factors and hyperfibrinolysis.
2. The concentration of NA correlates with thrombin formation and the correlation is stronger in higher doses of NA.
3. Thrombin formation will decrease more slowly in the group that will receive NA therapy in comparison to the group that will not receive NA therapy.

DETAILED DESCRIPTION:
STUDY DESIGN AND METHODS The research shall be carried out at the Department of Anaesthetics and Surgical Intensive Care/Intensive Care Unit (ICU) at the University Medical Centre Ljubljana and will begin once it is approved by the Slovenian National Medical Ethics Committee. Patients will be included in the research once the informed consent form is signed by their relatives or their legal guardian.

Patients and the course of the study The research study will focus on 60 consecutive patients with severe traumatic brain injury (TBI) hospitalised at the emergency unit's ICU, who will be treated according to the Advanced Trauma Life Support guidelines, will undergo a computerized tomography (CT) scan of the head, and will have been implanted with an electrode for monitoring intracranial pressure (ICP). Both female and male patients, age 18 to 80, with Glasgow Coma Scale (GCS) ≤ 8 and Head Abbreviated Injury Scale (AIS) ≥ 3 shall be included in the study. Patients with any kind of extracranial injury, patients receiving anticoagulation or anti aggregation therapy, patients with a known neurological, haematological, malign or liver disease, patients with an infection and after a cardiac arrest, after craniotomy, patients that have received transfusion of concentrated erythrocytes (> 1 bag) and/or fresh frozen plasma, thrombocyte plasma, patients with a body temperature of < 35°C and pregnant women will all be excluded from the study, as will be those cases where it will be impossible to perform targeted tests in the expected time frame.

At the ICU, patients will receive treatment according to the guidelines for the treatment of severe traumatic brain injury. All patients will be sedated with midazolam, they will receive analgesia with fentanyl, and when required considering the level of ICP, will also receive a 2% propofol infusion. They will all be mechanically ventilated. A non-heparinized central venous catheter and an artery catheter will both be routinely inserted in all cases. Blood samples for the study will be taken from the internal jugular vein with a singular puncture.

Systemic blood pressure, heart rate, central body temperature, peripheral blood oxygen saturation (SpO2), ICP, cerebral perfusion pressure (CPP) and bispectral index (BIS) of the depth of anaesthesia will be monitored at all times. Pupillary response and depth of sedation using the Richmond Agitation-Sedation Scale (RASS) will be performed once per hour. Hydration will be estimated with stroke volume variation (SVV) one or twice per day. Patients whose CPP will not meet the desired value (70 mmHg) will receive systemic intravenous infusion of NA solution (0.16 mg/ml) in the dosage required to meet the target CPP. Another CT scan will be performed 12 to 24 hours after injury and after sudden deterioration in health condition, if necessary.

Blood samples will be taken daily from the artery catheter to determine the values of electrolytes, glucose, number of leukocytes and haemogram, number of thrombocytes all of which are routinely performed on a daily basis.

In the periods of 1-3, 6, 12 and 24 hours after injury, a member of the research staff will collect a blood sample from the patient with a severe TBI via an arterial catheter in order to determine: the level of endogenous NA or of total, endogenous and exogenous NA, if the patient will have received continuous NA infusion, the number of thrombocytes, prothrombin time/international normalized ration (PT/INR), activated partial thromboplastin time (aPTT), fibrinogen, antithrombin (AT), D-dimer, rotational thromboelastometry (ROTEM) test results, platelet function with aggregometry (Multiplate), lactate level, pH balance, gas analysis (PaO2, PaCO2), HCO3, base deficit and arterial blood oxygen saturation (SaO2). Venipuncture shall be performed on patients with severe TBI in the periods of 1-3, 6, 12 and 24 hours after injury by a member of the research staff to collect a blood sample from the jugular vein in order to determine: the level of endogenous NA or of total, endogenous and exogenous NA, if the patient will have received continuous NA infusion, number of thrombocytes, PT/INR, aPTT, fibrinogen, tissue factor (TF), AT, thrombin-antithrombin complex (TAT); D-dimer, tissue-plasminogen activator antigen (t-PAAg), plasminogen activator inhibitor-1 antigen (PAI-1Ag), plasminogen activator inhibitor-1 activity (PAI-1Act), plasmin-antiplasmin complex (PAP), plasminogen activity; protein C antigen (PCAg), syndecan-1 (SDC-1), rotational thromboelastometry (ROTEM) test results, platelet function with aggregometry (Multiplate). In patients who will require an infusion of NA within 1-3 hours after hemostasis tests have already been taken, the NA level will be determine again 30 minutes after the infusion set, and all mentioned hemostasis tests from the internal jugular vein and arterial catheter will be re-controlled. CT will be repeated 12 and 24 hours after the injury and if necessary in the case of a sudden worsening of the clinical condition.

Patients with severe TBI will be divided into two groups. Group A for patients that will need an infusion of NA solution to meet the desired CPP, and Group B for patients that will not receive NA infusion. Group A will be further divided into three sub-groups: A1 for patients that will receive NA in the dose of 0.06-0.12 μg/kg/min, A2 for patients that will receive a dose of 0.13-0.2 μg/kg/min, and A3 for patients that will receive a dose of NA > 0.2 μg/kg/min. Absolute values of individual laboratory variables in different time intervals (1-3, 6, 12, 24 hours after injury) will be compared between Groups A and B, between sub-group A1 and B, A2 and B, and A3 and B; and between sub-groups A1, A2 and A3.

ELIGIBILITY:
Inclusion Criteria:

* patients with traumatic brain injury
* Glasgow Coma Scale ≤ 8
* Head Abbreviated Injury Scale (AIS) ≥ 3

Exclusion Criteria:

* patients with any kind of extracranial injury
* patients receiving anticoagulation or anti aggregation therapy
* patients with a known neurological disorders
* patients with haematological disorders
* patients with malign diseases
* patients with liver disease
* patients with any infection
* patients after cardiac arrest
* patients after craniotomy
* patients that have received transfusion of contentrated erythrocytes and/or fresh frozen plasma
* patients that have received thrombocyte plasma
* body temperature <35°C
* pregnant women

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The research study will focus on 60 consecutive patients with severe traumatic brain injury (TBI) hospitalised at the emergency unit's ICU at the University Medical Center Ljubljana, who will be treated according to the Advanced Trauma Life Support guidelines, will undergo a computerized tomography (CT) scan of the head, and will have been implanted with an electrode for monitoring intracranial pressure (ICP).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of noradrenalin plasma levels between group A and group B | 1 year
  Blood sempling from the internal jugular vein will be done after 3, 6, 12, 24 hours after the injury. Blood will be centrifugated and plasma extracted. Plasma will be sent in the central hospital laboratory for plasma noradrenalin concentration measurement. Concentration will be expressed in pg/ml.
Change of thrombin formation and fibrinolysis between group A and group B | 1 year
  Blood sempling from the internal jugular vein will be done after 3, 6, 12, 24 hours after the injury. Blood will be centrifugated and plasma extracted. Plasma will be sent in the central hospital laboratory for measurement of tissue factor concentration in mcg/ml, antithrombin concentration in percents and thrombin-antitrombin complex concentration, as indirect indicator of trombin generation (concentration will be expressed in ng/ml).
  Fibrinolysis will be measured by the plasma levels of D-dimer in mcg/L, tissue plasminogen activator antigen in mcg/ml, plasminogen activator inhibitor-1 antigen in IU/ml, plasminogen activator inhibitor activity in mcg/ml, plasmin antiplasmin complex in mcg/ml and plasminogen concentration in mcg/ml.

SECONDARY OUTCOMES:
Change in basic haemostasis test between two groups | 1 year
  Blood sempling from the internal jugular vein will be done after 3, 6, 12, 24 hours after the injury. Blood will be centrifugated and plasma extracted. Plasma will be sent in the central hospital laboratory. Change will be determinated by INR, activated partial trombin time in seconds, fibrinogen concentration in g/L and platelet count.
Change of syndecan-1 plasma level | 1 year
  Blood sempling from the internal jugular vein will be done after 3, 6, 12, 24 hours after the injury. Blood will be centrifugated and plasma extracted. Plasma will be sent in the central hospital laboratory. Change will be measured in ng/ml.
Change of protein-C antigen | 1 year
  Blood sempling from the internal jugular vein will be done after 3, 6, 12, 24 hours after the injury. Blood will be centrifugated and plasma extracted. Plasma will be sent in the central hospital laboratory. Concentration will be expressed in percentage.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stein SC, Smith DH. Coagulopathy in traumatic brain injury. Neurocrit Care. 2004;1(4):479-88. doi: 10.1385/NCC:1:4:479. PMID 16174954
- [Result] Pathak A, Dutta S, Marwaha N, Singh D, Varma N, Mathuriya SN. Change in tissue thromboplastin content of brain following trauma. Neurol India. 2005 Jun;53(2):178-82. doi: 10.4103/0028-3886.16404. PMID 16010055
- [Result] Laroche M, Kutcher ME, Huang MC, Cohen MJ, Manley GT. Coagulopathy after traumatic brain injury. Neurosurgery. 2012 Jun;70(6):1334-45. doi: 10.1227/NEU.0b013e31824d179b. PMID 22307074
- [Result] Stein SC, Graham DI, Chen XH, Smith DH. Association between intravascular microthrombosis and cerebral ischemia in traumatic brain injury. Neurosurgery. 2004 Mar;54(3):687-91; discussion 691. doi: 10.1227/01.neu.0000108641.98845.88. PMID 15028145
- [Result] Cohen MJ, Brohi K, Ganter MT, Manley GT, Mackersie RC, Pittet JF. Early coagulopathy after traumatic brain injury: the role of hypoperfusion and the protein C pathway. J Trauma. 2007 Dec;63(6):1254-61; discussion 1261-2. doi: 10.1097/TA.0b013e318156ee4c. PMID 18212647
- [Result] Rizoli SB, Jaja BN, Di Battista AP, Rhind SG, Neto AC, da Costa L, Inaba K, da Luz LT, Nascimento B, Perez A, Baker AJ, de Oliveira Manoel AL. Catecholamines as outcome markers in isolated traumatic brain injury: the COMA-TBI study. Crit Care. 2017 Feb 23;21(1):37. doi: 10.1186/s13054-017-1620-6. PMID 28228155
- [Result] Myburgh JA. Driving cerebral perfusion pressure with pressors: how, which, when? Crit Care Resusc. 2005 Sep;7(3):200-5. PMID 16545046
- [Result] Johansson PI, Stensballe J, Rasmussen LS, Ostrowski SR. A high admission syndecan-1 level, a marker of endothelial glycocalyx degradation, is associated with inflammation, protein C depletion, fibrinolysis, and increased mortality in trauma patients. Ann Surg. 2011 Aug;254(2):194-200. doi: 10.1097/SLA.0b013e318226113d. PMID 21772125
- [Result] von Kanel R, Heimgartner N, Stutz M, Zuccarella-Hackl C, Hansel A, Ehlert U, Wirtz PH. Prothrombotic response to norepinephrine infusion, mimicking norepinephrine stress-reactivity effects, is partly mediated by alpha-adrenergic mechanisms. Psychoneuroendocrinology. 2019 Jul;105:44-50. doi: 10.1016/j.psyneuen.2018.09.018. Epub 2018 Sep 14. PMID 30318393
- [Result] Tschuor C, Asmis LM, Lenzlinger PM, Tanner M, Harter L, Keel M, Stocker R, Stover JF. In vitro norepinephrine significantly activates isolated platelets from healthy volunteers and critically ill patients following severe traumatic brain injury. Crit Care. 2008;12(3):R80. doi: 10.1186/cc6931. Epub 2008 Jun 18. PMID 18564410